CLINICAL TRIAL: NCT01110681
Title: An Open, Non-comparative, Post-marketing, Multi-center Study to Evaluate Efficacy and Safety of SolestaTM for the Treatment of Fecal Incontinence
Brief Title: Study to Evaluate Solesta for Treatment of Fecal Incontinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 33DA0605, Q-Med AB
Record Dates: First submitted 2010-04-09; First posted 2010-04-27 (Estimated); Results first posted 2019-02-28 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2013-12

CONDITIONS: Fecal Incontinence
MeSH Terms: conditions — Fecal Incontinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Solesta (Experimental): Open label. Solesta (Dextranomer in gel of stabilized non-animal hyaluronate) The study treatment consisted of 4 submucosal injections, 1 mL Solesta each, in the proximal part of the high pressure zone in the anal canal.
  Re-treatment is allowed one month after initial treatment if the subject is still incontinent.
  Interventions: Device: Solesta (Dextranomer in gel of stabilized non-animal hyaluronate)

INTERVENTIONS:
Device: Solesta (Dextranomer in gel of stabilized non-animal hyaluronate)
  Other Names: Solesta

SUMMARY:
The study will evaluate the safety and efficacy of Solesta as an injectable bulking agent in the treatment of fecal incontinence for a total of 24 months after completed treatment.

ELIGIBILITY:
Inclusion Criteria:

* 18-80 years of age, male or female
* Screening fecal incontinence severity score (CCFIS)
* Fecal incontinence episodes over a 28-day period
* Failed conservative treatment for fecal incontinence

Exclusion Criteria:

* Complete external sphincter disruption
* Significant anorectal disease
* Anorectal surgery within the last 12 months prior to the study
* Active Inflammatory Bowel Disease
* Immunodeficiency or receiving immunosuppressive therapy
* Malignancies in remission for less than 1 years prior to the study
* Bleeding disorders or receiving anticoagulant therapy
* Chemotherapy within the last 6 months prior to the study
* Prior Pelvic radiotherapy
* Pregnant or breast-feeding women, or women of childbearing potential not practicing adequate contraception or planning to stop such contraception within the first year of the study
* Women within 6 months post partum
* Participation in any other clinical study within 3 month prior to the study
* Other severe conditions or in other ways unsuitable to participate according to investigator judgement

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2007-11; Primary Completion 2009-11 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Head of Medical Affairs Q-Med AB, Study Director — Galderma R&D; Tom Oresland, MD, Principal Investigator — Akershus University Hospital, Lorenskog, Norway
Locations (15):
- St. Paul's Hospital, Vancouver, Canada
- Helsingin yliopistollinen keskussairaala, HUS, Finland
- France (3):
  - CHU-Hotel-Dieu, Nantes
  - Hôpital Saint Joseph, Paris
  - CHU de Rouen 1 rue Germont service de chirurgie et digestive, Rouen
- Germany (3):
  - Koloproktologische Praxis, Kiel
  - Klinik für Allgemein- und Vizeralchirurgie, Ludwigsburg
  - Enddarmzentrum Mannheim, Mannheim
- Italy (3):
  - University of Bari - Coloproctological Unit of Bari Policinico di Bari Piazza, Bari
  - Univ. degli Studi di Padova Hospital Clinica Chirurgica, Padua
  - Policlinico Umberto I, Rome
- Akershus universitetssykehus, Nordbyhagen, Norway
- Spain (3):
  - Hospital Clinic Provincial, Barcelona
  - Hospital Juan Ramón Jiménez, Huelva
  - Hospital General Univ. de Valéncia, Valencia

RESULTS

PARTICIPANT FLOW:
Groups:
- Solesta: Open label.
  Solesta (Dextranomer in gel of stabilized non-animal hyaluronate) : Submucosal injections. Re-treatment is allowed one month after initial treatment if the subject is still incontinent.
Period: Overall Study
Arm/Group | Solesta
Started | 115
Completed | 83
Not Completed | 32

BASELINE CHARACTERISTICS:
Arm/Group | Solesta
Number analyzed (Participants) | 115
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.5 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 100
  Male | 15
Region of Enrollment [Number; unit: participants]
  France | 23
  Canada | 12
  Finland | 10
  Spain | 16
  Norway | 3
  Germany | 21
  Italy | 30

OUTCOME MEASURES:

1. Primary Outcome: Responder Rate in Number of Fecal Incontinence Episodes
Description: Responder rate in number of fecal incontinence episodes change from baseline at 12 month.
  Defined as responders at 12 month after treatment. A responder was defined as 50% or more reduction in the number of fecal incontinence episodes (28-day diary data)of solid or loose stool, compared to baseline.
Time Frame: 12 months after last treatment compared to baseline
Population: Intention to treat (all subjects who were treated with study product). Primary analysis were based on observed data. A Last-Observation-Carried -Forward (LOCF) technique was also used where the last performed efficacy assessment was carried forward to impute any subsequent missing values.
Measure: Number (95% Confidence Interval); unit: percentage of responders
Arm/Group | Solesta
Number analyzed (Participants) | 87
percentage of responders | 64.4 [54.3 to 74.4]

2. Secondary Outcome: Number of Fecal Incontinence Episodes.
Description: Number of fecal incontinence episodes, change from baseline (change in patient diary data at 12 month).
Time Frame: at 12 month - change from baseline
Population: as for outcome 1
Measure: Mean (Full Range); unit: episodes
Arm/Group | Solesta
Number analyzed (Participants) | 88
episodes | -10.94 [-82.2 to 45.6]

3. Secondary Outcome: Fecal Incontinence Severity Using the Cleveland Clinic Florida Incontinence Score
Description: Cleveland Clinic Florida Incontinence Score (CCFIS) is a composite score of incontinence severity that measures the frequencies of gas leakage, leakage of solid or loose stool, use of protective pads and lifestyle alterations. The score ranges from 0 (representing complete continence)to 20 (representing complete incontinence).
  Change from baseline.
Time Frame: 12 month - change from baseline
Population: Intention to treat. Primary analysis were based on observed data. A Last-Observation-Carried -Forward (LOCF) technique was also used where the last performed efficacy assessment was carried forward to impute any subsequent missing values.
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Solesta
Number analyzed (Participants) | 90
units on a scale | -4.79 [-18.0 to 5.0]

4. Secondary Outcome: Fecal Incontinence Quality of Life (FIQL)
Description: Fecal Incontinence Quality of Life is a disease specific questionnaire composed of a total of 29 questions questions divided into four domains: Lifestyle, Coping/Behavior, Depression/Self perception, and Embarrassment. The FIQL mean score ranges from 1 to 4 for the Lifestyle, Coping/Behavior and Embarrassment domains, and from 1 to 4.429 for Depression/Self-Perception domain. Mean score were calculated for each of the four domains. The more the subject is affected by fecal incontinence the lower value. Change from baseline.
Time Frame: At 12 month - change from baseline
Population: as for outcome 3
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Solesta
Number analyzed (Participants) | 77
score on a scale
  Lifestyle | 0.49 [-1.3 to 2.9]
  Coping/behaviour | 0.66 [-1.2 to 3.0]
  Depression/Self perception | 0.52 [-2.5 to 3.0]
  Embarrassment | 0.78 [-1.7 to 3.0]

5. Secondary Outcome: Number of Incontinence-free Days
Description: Number of incontinence-free days, change from baseline (change in patient diary data at 12 month).
Time Frame: At 12 month- change from baseline
Population: as for outcome 1
Measure: Mean (Full Range); unit: days
Arm/Group | Solesta
Number analyzed (Participants) | 88
days | 7.1 [-21.5 to 28]

ADVERSE EVENTS:
Arm/Group | Solesta
Serious Adverse Events (participants affected / at risk) | 19/115
Other Adverse Events (participants affected / at risk) | 20/115
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Solesta (N=115)
Perineal abscess (Infections and infestations) | 1 (1)
Rectovaginal septum abscess (Infections and infestations) | 1 (1)
Rectal abscess (Infections and infestations) | 1 (1)
Rectal prolapse (Gastrointestinal disorders) | 2 (2)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (3)
Proctalgia (Gastrointestinal disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Breast infection (Infections and infestations) | 1 (1)
Cardiac failure acute (Cardiac disorders) | 1 (2)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Fecal incontinence (Gastrointestinal disorders) | 1 (1)
Gastroenteritis (Gastrointestinal disorders) | 1 (1)
Hemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 (1)
Hypothyriodism (Endocrine disorders) | 1 (1)
Polycystic liver disease (Hepatobiliary disorders) | 1 (1)
Postmenopausal hemorrhage (Reproductive system and breast disorders) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1)
Sjögrens syndrome (Immune system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Solesta (N=115)
Proctalgia (Gastrointestinal disorders) | 15 (15)
Pyrexia (General disorders) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less